CLINICAL TRIAL: NCT00124865
Title: Safety and Immunogenicity Evaluation of an Intranasal Recombinant Flagellin Subunit Campylobacter Vaccine (rFla-MBP) in Volunteers
Brief Title: Intranasal Recombinant Flagellin Subunit Campylobacter Vaccine (rFla-MBP) Dose-Ranging Study
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NMRC 2002.0003; WRAIR 949 (Other: WRAIR); HSRRB A-11697 (Other: USAMRMC); rFla-MBP (Other: NMRC)
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Diarrhea
Keywords: Campylobacter; Bacterial enteritis
MeSH Terms: conditions — Diarrhea

INTERVENTIONS:
Biological: rFla-MBP

SUMMARY:
This study is an open-labeled dose escalating trial in which a total of 32 subjects will receive one of four intranasal rFla-MBP vaccine doses.

DETAILED DESCRIPTION:
This is an open labeled dose escalating trial in which a total of 32 subjects will receive one of four intranasal rFla-MBP vaccine doses according to the following chart:

Group / N* / rFla-MBP

A / 8/ 25 micrograms

B / 8/ 125 micrograms

C / 8/ 625 micrograms

D / 8/ 1000 micrograms

* minimum of 6 volunteers per group

An interval no less than 60 days following the first dose will separate the first dose of each volunteer group receiving different rFla-MBP doses. All volunteers will receive three immunizations. The first dosing time point is Day 0, the second is Day 14 (+/- 1 day), the third is day 28 (+/- 2 days). Blood and stool specimens will be collected at intervals to examine systemic and mucosal vaccine antigen-specific immune responses. Vaccine safety will be actively monitored during vaccination and for 28 days following the third vaccine dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* 70% accuracy on comprehension test
* Availability for required visits and telephone follow up

Exclusion Criteria:

* Pregnancy or breastfeeding
* Chronic health problems
* Abnormalities found on physical examination
* Use of immunosuppressive drugs, such as corticosteroids or chemotherapy
* Positive blood test for HIV-1, hepatits B surface antigen (HBsAG) or hepatitis C virus (HCV)
* Abnormalities found on basic laboratory screening
* Prior exposure to Campylobacter
* Current smoker
* Chronic sinusitis or seasonal rhinitis

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-07; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Local and systemic reactions
Mucosal immunogenicity
Systemic immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: David Tribble, MD, DrPH, Principal Investigator — Naval Medical Research Center
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States